CLINICAL TRIAL: NCT06756984
Title: A Prospective Cohort Study on the Long-Term Outcomes and Prognostic Factors of Different Surgical Techniques for the Treatment of Sacral Tarlov Cysts
Brief Title: Long-Term Outcomes of Different Surgical Techniques for Sacral Tarlov Cysts: A Prospective Cohort Study
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Jishuitan Hospital (Other)
Responsible Party: Principal Investigator, Liu longqi, MSc, Neurosurgeon, Department of Neurosurgery, Beijing Jishuitan Hospital, Beijing Jishuitan Hospital
Other Study IDs: STC_2025
Record Dates: First submitted 2024-12-24; First posted 2025-01-03 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Sacral Tarlov Cysts; Symptomatic Sacral Cysts; Chronic Pain Related to Sacral Cysts; Neurological Dysfunction Associated With Tarlov Cysts
MeSH Terms: conditions — Tarlov Cysts | interventions — Plastic Surgery Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Partial Cyst Wall Resection with Nerve Root Sleeve Plasty: Participants in this group will undergo partial resection of the cyst wall combined with nerve root sleeve plasty. This technique involves reducing the cyst size and reconstructing the nerve root sleeve to restore nerve function and reduce symptoms.
  Interventions: Procedure: Partial Cyst Wall Resection with Nerve Root Sleeve Plasty
- Partial Cyst Wall Resection with Nerve Root Sleeve Reinforcement and Reconstruction: Participants in this group will undergo partial resection of the cyst wall along with reinforcement and reconstruction of the nerve root sleeve. This method provides additional structural stability to the nerve root and aims to reduce the risk of recurrence and improve postoperative outcomes.
  Interventions: Procedure: Partial Cyst Wall Resection with Nerve Root Sleeve Reinforcement and Reconstruction:
- Autologous Fat/Muscle with Fibrin Glue Microscopic Cyst Filling: Participants in this group will receive autologous fat or muscle tissue filling of the cyst cavity combined with fibrin glue sealing under microscopic guidance. This technique aims to obliterate the cyst cavity, prevent cerebrospinal fluid leakage, and enhance symptom relief and recovery.
  Interventions: Procedure: Autologous Fat/Muscle with Fibrin Glue Microscopic Cyst Filling

INTERVENTIONS:
Procedure: Partial Cyst Wall Resection with Nerve Root Sleeve Plasty — Surgical technique involving partial removal of the cyst wall to decompress the nerve root, followed by plasty of the nerve root sleeve to restore nerve function and prevent recurrence.
  Groups: Partial Cyst Wall Resection with Nerve Root Sleeve Plasty
Procedure: Partial Cyst Wall Resection with Nerve Root Sleeve Reinforcement and Reconstruction: — Advanced surgical technique combining partial cyst wall removal with additional reinforcement and reconstruction of the nerve root sleeve to provide enhanced support and reduce the risk of cyst recurrence.
  Groups: Partial Cyst Wall Resection with Nerve Root Sleeve Reinforcement and Reconstruction
Procedure: Autologous Fat/Muscle with Fibrin Glue Microscopic Cyst Filling — Minimally invasive surgical technique where autologous fat or muscle tissue is used to fill the cyst cavity, and fibrin glue is applied to seal the defect, aiming to obliterate the cyst and prevent cerebrospinal fluid leakage.
  Groups: Autologous Fat/Muscle with Fibrin Glue Microscopic Cyst Filling

SUMMARY:
Brief Summary

The goal of this observational study is to evaluate the long-term outcomes of different surgical techniques for sacral Tarlov cysts in adult patients aged 18-75 years diagnosed with symptomatic sacral Tarlov cysts. The main questions it aims to answer are:

* Does one surgical technique result in better pain relief (measured by VAS score) and functional recovery (measured by JOA score) compared to others?
* How do different surgical techniques impact the long-term recurrence rate and complication rate?

Researchers will compare three surgical techniques:

1. Partial cyst wall resection with nerve root sleeve plasty.
2. Partial cyst wall resection with nerve root sleeve reinforcement and reconstruction.
3. Autologous fat/muscle with fibrin glue microscopic cyst filling.

Participants will:

* Undergo one of the three surgical procedures based on clinical indications.
* Complete preoperative and postoperative assessments, including pain and functional scoring, as well as MRI evaluations at baseline and during follow-up.
* Participate in a follow-up program for up to 2 years to monitor outcomes and recurrence.

ELIGIBILITY:
Inclusion Criteria

1. Age 18-75 years.
2. Diagnosed with symptomatic sacral Tarlov cysts confirmed by MRI.
3. Presence of at least one of the following symptoms:

   * Persistent sacral or lower back pain (VAS score ≥ 4).
   * Neurological deficits such as lower extremity numbness or weakness.
   * Bowel, bladder, or sexual dysfunction attributable to the cyst.
4. Eligible for surgical intervention based on clinical evaluation.
5. Willing and able to provide written informed consent.

Exclusion Criteria

1. History of prior sacral Tarlov cyst surgery.
2. Concurrent spinal conditions requiring separate surgical intervention.
3. Active infection or systemic inflammatory disease.
4. Severe comorbidities that increase surgical risk (e.g., advanced cardiac or pulmonary disease).
5. Pregnancy or lactation.
6. Inability to comply with follow-up requirements.
7. Known allergy or contraindication to surgical materials (e.g., fibrin glue).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adult patients aged 18-75 years diagnosed with symptomatic sacral Tarlov cysts, recruited from the Department of Neurosurgery at Beijing Jishuitan Hospital. Participants must exhibit persistent symptoms such as sacral or lower back pain, neurological deficits (e.g., numbness or weakness in the lower extremities), or bowel/bladder/sexual dysfunction attributable to the cyst, confirmed by MRI. The study focuses on individuals eligible for surgical intervention without significant comorbidities or prior related surgeries. This population represents a clinically relevant cohort for evaluating the efficacy and safety of different surgical techniques for sacral Tarlov cysts.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-05-13 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain Reduction Assessed by Visual Analog Scale (VAS) | Baseline, 1 month, 3 months, 6 months, 12 months and 24 months postoperatively
Neurological Function Improvement Assessed by Japanese Orthopedic Association (JOA) Score | Baseline, 1 month, 3 months, 6 months, 12 months and 24 months postoperatively

SECONDARY OUTCOMES:
Recurrence Rate of Sacral Tarlov Cysts | 12 months postoperatively and annually up to 2 years

IPD SHARING:
Plan to Share IPD: No